CLINICAL TRIAL: NCT06962020
Title: Selection and Efficacy-Influencing Factors of First-Line Biologic Agents in Moderate-to-Severe Ulcerative Colitis: A Prospective, Multi-Center, Real-World Study
Brief Title: Selection and Efficacy-Influencing Factors of First-Line Biologic Agents in Moderate-to-Severe Ulcerative Colitis
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Clinical Professor, Xijing Hospital of Digestive Diseases
Other Study IDs: KY20232425-F-1
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis (UC)
Keywords: biologics; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The IFX group: The first-line use of IFX group regularly uses IFX treatment for 3 cycles before continuing to use IFX or adjusting to VDZ treatment.
  Interventions: Drug: first-line biologic：IFX
- The VDZ group: The first-line use of VDZ group regularly uses VDZ treatment for 3 cycles before continuing to use VDZ or adjusting to IFX treatment.
  Interventions: Drug: first-line biologic:VDZ

INTERVENTIONS:
Drug: first-line biologic：IFX — IFX is administered intravenously at a dose of 5-10mg/kg, once at weeks 0, 2, and 6 (or 0, 1, and 5), and then every 8 weeks at a dose of 5mg/kg for maintenance treatment. VDZ is administered intravenously at a dose of 300mg/time, once at weeks 0, 2, and 6, and then every 8 weeks at a dose of 300mg for maintenance treatment.
  Groups: The IFX group
Drug: first-line biologic:VDZ — IFX is administered intravenously at a dose of 5-10mg/kg, once at weeks 0, 2, and 6 (or 0, 1, and 5), and then every 8 weeks at a dose of 5mg/kg for maintenance treatment. VDZ is administered intravenously at a dose of 300mg/time, once at weeks 0, 2, and 6, and then every 8 weeks at a dose of 300mg for maintenance treatment.
  Groups: The VDZ group

SUMMARY:
The purpose of this prospective, multicenter, real-world study is to compare the efficacy differences and influencing factors of different first-line biologics in patients with moderate to severe ulcerative colitis. The question that this study aims to answer is: When treating patients with moderate to severe ulcerative colitis, should IFX or VDZ be prioritized as the first-line choice for biologics?, Which biological agent has better therapeutic effect?. Researchers will observe and follow up with patients with moderate to severe ulcerative colitis treated with different biologics on the front line, evaluate their condition changes, eliminate relevant interfering factors, and draw the final conclusion.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18-70 years old, gender not limited;
* According to international guidelines and consensus, patients with ulcerative colitis should be diagnosed to exclude radiation enteritis, infectious enteritis, tumor related diseases, etc;
* Patients assessed as moderate to severe ulcerative colitis based on the Mayo score;
* During the follow-up period, no relevant treatments (drugs and surgery) were used that could affect the assessment of the efficacy of biologics

Exclusion Criteria:

* Patients with hemodynamic instability;
* Patients with obvious liver and kidney function injury: bilirubin, aminotransferase (ALT, AST) exceeded the upper limit of normal by 2 times; eGFR<60ml/min or dialysis patients;
* Patients allergic to IFX or VDZ;
* Patients whose primary disease was gastrointestinal malignancy;
* Patients currently suffering from serious or uncontrolled underlying diseases of the blood, digestive tract, metabolism, endocrine, lung, heart, nervous system, mental system, etc.;
* Female patients during pregnancy and breastfeeding (including patients with reproductive needs);
* Patients with current infection with infectious diseases (hepatitis B, hepatitis C, syphilis, AIDS, tuberculosis, etc.);
* Patients who cannot cooperate with regular follow-up and review of laboratory indicators;
* Any other circumstances which, in the opinion of the investigator, would render the subject unfit for study inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to severe UC patients treated with biological agents in the Xijing Hospital of Digestive Diseases
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rates and endoscopic remission rates at 14 weeks, 30 weeks, 52 weeks, and 2 years after first-line biologics treatment | From enrollment to the end of treatment at 2 years.
  Evaluate the clinical remission rate and endoscopic remission rate of first-line biologics treatment at 14 weeks, 30 weeks, 52 weeks, and 2 years based on the Mayo scoring system and endoscopic examination results

SECONDARY OUTCOMES:
Clinical response rate, endoscopic response rate, and hormone free response rate at 14 weeks, 30 weeks, 52 weeks, and 2 years after first-line biologics treatment | From enrollment to the end of treatment at 2 years.
  Evaluate the clinical response rate, endoscopic response rate, and hormone free response rate at 14 weeks, 30 weeks, 52 weeks, and 2 years after first-line biologic therapy based on the Mayo scoring system and endoscopic examination results
Factors affecting the efficacy of two biological agents in the treatment process | From enrollment to the end of treatment at 2 years.
  After balancing confounding factors through PSM, IPTW, and other methods, the factors affecting the efficacy of biologics were analyzed through survival analysis curves

CONTACTS AND LOCATIONS:
Overall Officials: Min Chen, Study Director — Xijing Hospital of Digestive Diseases
Locations (1):
- Xijing Hospital of Digestive Diseases, Shanxi, Xi'an, China

IPD SHARING:
Plan to Share IPD: No